CLINICAL TRIAL: NCT00559403
Title: South African Adolescent Health Promotion Project
Brief Title: Effect of HIV/STD Risk Reduction Program on South African Adolescents
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, John Jemmott, Kenneth B. Clark Professor of Communication and Psychiatry, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: R01MH065867 (NIH); R01MH065867 (NIH); DAHBR AZ-A (Other: National Institute of Mental Health)
Record Dates: First submitted 2007-11-14; First posted 2007-11-16 (Estimated); Last update posted 2015-09-25 (Estimated); Status verified 2015-09

CONDITIONS: HIV Infections; Sexually Transmitted Disease
Keywords: Human immunodeficiency virus; South Africa; Intervention Studies; Sexual Behavior; Adolescents; STD; HIV Seronegativity
MeSH Terms: conditions — HIV Infections; Sexually Transmitted Diseases; Acquired Immunodeficiency Syndrome; Sexual Behavior | interventions — Health Promotion

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- HIV/STD Sessions (Experimental): The HIV/STD Risk-Reduction Intervention arm focuses on reducing the risk of STDs, including HIV.
  Interventions: Behavioral: HIV/STD Risk-Reduction
- Health Promotion Control Sessions (Active Comparator): The Health Promotion Intervention arm focuses on physical activity, diet, and other behaviors linked to risk of heart disease, high blood pressure, stroke, diabetes, and certain cancers, which are all leading causes of morbidity and mortality among South Africans.
  Interventions: Behavioral: Health Promotion

INTERVENTIONS:
Behavioral: HIV/STD Risk-Reduction — Let Us Protect Our Future consists of twelve 1-hour sessions to increase knowledge, motivation, and skills in practicing abstinence and condom use. It is highly structured, and Xhosa-speaking male and female co-facilitators implement the program using standardized manuals. Treatment sessions include mixed-gender and single-gender activities, games, brainstorming, and role-playing. Comic workbooks are used to address abstinence, condom use, and how risky behavior affects goals and dreams. The Xhosa culture is taken into account, including cultural transformations in urban township settings. Take-home assignments enlist parents' help to empower their children to reduce their STD risk and ensure that parents are aware of the nature of the treatment program.
  Other Names: Let Us Protect Our Future
  Arms: HIV/STD Sessions
Behavioral: Health Promotion — The health promotion treatment is structurally similar to the HIV/STD treatment: each has the same number of sessions and sessions led by Xhosa-speaking male and female co-facilitators. It focuses on behaviors linked with risk of heart disease, diabetes, high blood pressure, certain cancers, and alcohol and drug abuse, which are all leading causes of morbidity and mortality among South Africans. Participants are taught that healthful behaviors, including eating habits, physical activity, dental hygiene, and avoidance of cigarette smoking and substance use, can prevent these health problems. Comic workbook story lines are used to increase risk perception and awareness of health risks. Take-home assignments are used to foster communication with parents about healthful lifestyle.
  Arms: Health Promotion Control Sessions

SUMMARY:
This study will evaluate the effect of an HIV/STD risk-reduction program on the sexual behavior of South African adolescents.

DETAILED DESCRIPTION:
HIV is a virus that can lead to acquired immunodeficiency syndrome (AIDS), a disease that breaks down the immune system and allows for entry of life-threatening secondary infections. HIV is transmitted through the exchange of bodily fluids, primarily through sexual intercourse. South Africa has been one of the countries in which the AIDS pandemic has had an especially devastating effect. New cases of HIV infection in South Africa have been occurring at a high rate in people 15 to 24 years of age. There is no vaccine or cure for HIV yet, making disease prevention methods imperative. An important part of the prevention process is early education on HIV to reduce sexual-risk behavior and to promote safe sexual practices. This study will evaluate the effect of an HIV/STD risk-reduction program on the sexual behavior of South African adolescents.

In this single-blind study, participants will include sixth grade students from 18 South African schools that meet study criteria. The participants will be randomly divided into 2 structurally similar treatment groups. One group will take part in HIV/STD risk-reduction sessions, while the other group will take part in health promotion sessions. There will be 12 total sessions, each lasting 1 hour. The participants in the HIV/STD risk-reduction group will be taught to practice abstinence and condom use through interactive activities, comic workbooks, and take-home assignments. Through similar methods, the participants in the health promotion group will be taught about general health problems, such as heart disease, diabetes, alcohol and drug abuse, and certain cancers. Participants will also be taught healthful behaviors to help prevent these health problems. All participants will provide self-reports of sexual behavior and precautionary methods used in sexual intercourse immediately before the first and after the last treatment sessions. Follow-up evaluations will occur at Months 3, 6, 12, 42, and 54 months post-treatment. STDs will be assessed 42 and 54 months post-treatment

ELIGIBILITY:
Inclusion Criteria:

* Schools, with Grade 6 learners, that served the general population of learners, not just those with learning disabilities
* Grade 6 learners at participating schools with signed parent/guardian consent forms

Exclusion Criteria:

* Schools exclusively serving children with learning disabilities

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1057 (Actual)
Dates: Start 2004-10; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Protection use in sexual intercourse | Measured at Month 12

SECONDARY OUTCOMES:
Sexual intercourse considerations: number of sexual partners, sexual debut, anal intercourse, consistency of condom use | Measured at Month 12
Theoretical mediators of abstinence (e.g., self-efficacy to avoid having sexual intercourse) | Measured at Month 12
Theoretical mediators of condom use (e.g., self-efficacy to use condoms) | Measured at Month 12
HIV/STD risk-reduction knowledge | Measured at Month 12
Condom-use knowledge | Measured at Month 12
Biologically confirmed STDs | Measured at Month 42
  Positive test for chlamydial infection, gonorrhea, and trichomoniasis

CONTACTS AND LOCATIONS:
Overall Officials: John B. Jemmott III, PhD, Principal Investigator — University of Pennsylvania

REFERENCES:
- [Background] Jemmott LS, Jemmott JB 3rd, Ngwane Z, Icard L, O'Leary A, Gueits L, Brawner B. 'Let Us Protect Our Future' a culturally congruent evidenced-based HIV/STD risk-reduction intervention for young South African adolescents. Health Educ Res. 2014 Feb;29(1):166-81. doi: 10.1093/her/cyt072. Epub 2013 Aug 20. PMID 23962491
- [Background] Jemmott JB 3rd, Heeren GA, Ngwane Z, Hewitt N, Jemmott LS, Shell R, O'leary A. Theory of planned behaviour predictors of intention to use condoms among Xhosa adolescents in South Africa. AIDS Care. 2007 May;19(5):677-84. doi: 10.1080/09540120601084308. PMID 17505930
- [Result] Jemmott JB 3rd, Jemmott LS, O'Leary A, Ngwane Z, Lewis DA, Bellamy SL, Icard LD, Carty C, Heeren GA, Tyler JC, Makiwane MB, Teitelman A. HIV/STI risk-reduction intervention efficacy with South African adolescents over 54 months. Health Psychol. 2015 Jun;34(6):610-21. doi: 10.1037/hea0000140. Epub 2014 Aug 11. PMID 25110841
- [Result] O'Leary A, Jemmott JB 3rd, Jemmott LS, Bellamy S, Ngwane Z, Icard L, Gueits L. Moderation and mediation of an effective HIV risk-reduction intervention for South African adolescents. Ann Behav Med. 2012 Oct;44(2):181-91. doi: 10.1007/s12160-012-9375-4. PMID 22618963
- [Result] Jemmott JB 3rd, Jemmott LS, O'Leary A, Ngwane Z, Icard LD, Bellamy SL, Jones SF, Landis JR, Heeren GA, Tyler JC, Makiwane MB. School-based randomized controlled trial of an HIV/STD risk-reduction intervention for South African adolescents. Arch Pediatr Adolesc Med. 2010 Oct;164(10):923-9. doi: 10.1001/archpediatrics.2010.176. PMID 20921349
- [Result] Jemmott JB 3rd, Jemmott LS, O'Leary A, Ngwane Z, Icard L, Bellamy S, Jones S, Landis JR, Heeren GA, Tyler JC, Makiwane MB. Cognitive-behavioural health-promotion intervention increases fruit and vegetable consumption and physical activity among South African adolescents: a cluster-randomised controlled trial. Psychol Health. 2011 Feb;26(2):167-85. doi: 10.1080/08870446.2011.531573. PMID 21318928
- [Result] O'Leary A, Jemmott JB 3rd, Jemmott LS, Teitelman A, Heeren GA, Ngwane Z, Icard LD, Lewis DA. Associations between psychosocial factors and incidence of sexually transmitted disease among South African adolescents. Sex Transm Dis. 2015 Mar;42(3):135-9. doi: 10.1097/OLQ.0000000000000247. PMID 25668645
- [Derived] Jemmott JB 3rd, O'Leary A, Jemmott LS, Ngwane ZP, Teitelman AM, Makiwane MB, Bellamy SL. Effect of a Behavioral Intervention on Perpetrating and Experiencing Forced Sex Among South African Adolescents: A Secondary Analysis of a Cluster Randomized Trial. JAMA Netw Open. 2018 Aug 3;1(4):e181213. doi: 10.1001/jamanetworkopen.2018.1213. PMID 30646113